CLINICAL TRIAL: NCT06652464
Title: The Relationship Between Maresin-1 and Resolvin-D1 Levels and Disease Activity in Ulcerative Colitis
Brief Title: Maresin-1 and Resolvin-D1 Levels and Disease Activity in Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, selim demirci, Principal Investigator, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2024 - 01/07
Record Dates: First submitted 2024-10-15; First posted 2024-10-22 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Disease Activity; Remission of Ulcerative Colitis; Ulcerative Colitis Flare
Keywords: maresin-1; resolvin-D1; ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Active: Group of ulcerative colitis patients considered active according to the Mayo score. (30 patients)
- Remission: Group of ulcerative colitis patients considered remission according to the Mayo score. (30 patients)
- Control: Group without ulcerative colitis or inflammatory disease. (30 patients)

SUMMARY:
Specialized pro-resolving mediators (SPMs), which are typically thought to be formed via consecutive steps of oxidation of polyenoic fatty acids, have been shown to suppress inflammation and promote timely resolution of inflammation. They are mainly divided into four categories: lipoxins, resolvins, protectins, and maresins. The study will compare Maresin-1 and Resolvin-D1 levels in ulcerative colitis patients with those in the control group.

DETAILED DESCRIPTION:
Ulcerative colitis is a chronic inflammatory bowel disease characterized by inflammation of the superficial colonic mucosa, which starts in the rectum and diffusely extends throughout the colon, with alternating periods of flare-ups and remission. The diagnosis, activity, and treatment outcomes of ulcerative colitis are evaluated through a combination of symptoms, clinical examination, laboratory tests, radiology, endoscopy, and histological findings. Assessing inflammatory activity is crucial for approaching the disease and shaping treatment. Therefore, studies have aimed to identify the ideal disease marker. In recent years, there has been a search for non-invasive, easy, and quick laboratory markers to evaluate disease activity and treatment response. The optimal marker should be disease-specific, accurately reflect disease activity, be easily applicable in clinical practice, and identify patients at risk of relapse. Many clinical activity indicators and non-invasive markers have been used for this purpose, but they have only provided indirect findings in assessing disease activity.

When the impact of inflammation reaches a certain stage, a number of endogenous pro-resolving lipid mediators are synthesized to promote the resolution of inflammation. These mediators remove pro-inflammatory mediators and inflammatory cells from the site, repair damaged tissues, and eventually terminate inflammatory responses. If they cannot be produced at adequate levels and/or fail to function properly, inflammation cannot resolve during this process, leading to a chronic inflammatory phase. Several endogenous pro-resolving lipid mediators such as maresins, lipoxins, protectins, and resolvins have been discovered in recent years through scientific research. Many studies in the literature indicate that these mediators maintain a balance of pro-inflammatory chemical mediators, reduce the tissue infiltration of PMNLs (polymorphonuclear leukocytes), enhance macrophage efferocytosis and phagocytosis, and decrease collateral tissue damage caused by phagocytic cells.

Maresin-1 and resolvin-D1 are lipid molecules synthesized in macrophages and are produced from omega-3 polyunsaturated fatty acid, docosahexaenoic acid (DHA), and have been identified as a novel type of inflammatory mediator. Multiple studies have shown that Maresin-1 can control the inflammatory response by inhibiting neutrophil infiltration, downregulating the production of pro-inflammatory mediators, inhibiting NF-κB activation, restoring the Treg/Th17 balance, and alleviating endoplasmic reticulum stress.

Resolvin-D1 and Maresin-1 exhibit anti-inflammatory activity.The study aims to compare the serum levels of Resolvin-D1 (RvD1) and Maresin-1 (Mar1) during remission and active phases of ulcerative colitis with those in a control group, to evaluate whether they correlate with clinical and laboratory features, and to determine their potential use as markers reflecting inflammation in the diagnosis of ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

• Patients with ulcerative colitis in active and remission phases, and a control group without acute or chronic inflammatory disease.

Exclusion Criteria:

* Active malignancy
* Chronic kidney disease
* Diabetes mellitus
* Collagen tissue disease
* History of colectomy
* Acute infection
* Pregnancy / lactation period
* Within the past week, history of omega-3 dietary supplementation, non-steroidal anti-inflammatory drug use, or fish consumption.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with active and remission phase ulcerative colitis and those in the control group who presented to the gastroenterology outpatient clinic of our hospital.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
İnflammatory markers | Up to 2 months
  Maresin-1 and Resolvin-D1 levels in study groups

SECONDARY OUTCOMES:
İnflammatory markers | Up to 2 months
  White blood cell and CRP levels in study groups.

CONTACTS AND LOCATIONS:
Overall Officials: selim demirci, medical doctor, Principal Investigator — Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Locations (1):
- Abdurrahman Yurtaslan Oncology and Training Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serhan CN, Savill J. Resolution of inflammation: the beginning programs the end. Nat Immunol. 2005 Dec;6(12):1191-7. doi: 10.1038/ni1276. PMID 16369558
- [Background] Buckley CD, Gilroy DW, Serhan CN. Proresolving lipid mediators and mechanisms in the resolution of acute inflammation. Immunity. 2014 Mar 20;40(3):315-27. doi: 10.1016/j.immuni.2014.02.009. PMID 24656045
- [Background] Serhan CN, Yang R, Martinod K, Kasuga K, Pillai PS, Porter TF, Oh SF, Spite M. Maresins: novel macrophage mediators with potent antiinflammatory and proresolving actions. J Exp Med. 2009 Jan 16;206(1):15-23. doi: 10.1084/jem.20081880. Epub 2008 Dec 22. PMID 19103881